CLINICAL TRIAL: NCT06866574
Title: A Multicenter, Randomized, Double-Blind, Aluminum Adjuvant-Controlled Phase III Clinical Trial to Evaluate the Efficacy, Immunogenicity, and Safety of a Recombinant Human Papillomavirus 9-Valent (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) Vaccine (E. Coli) in Chinese Males Aged 18 to 45 Years
Brief Title: A Phase III Trial to Evaluate the Efficacy, Immunogenicity and Safety of a Recombinant Human Papillomavirus 9-Valent (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) Vaccine (E.Coli) in Chinese Males
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xiamen University (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry)
Responsible Party: Principal Investigator, Jun Zhang, Professor, Xiamen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HPV-PRO-015
Record Dates: First submitted 2025-02-27; First posted 2025-03-10 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Penile/Perineal /Perianal Intraepithelial Neoplasia; Anal Intraepithelial Neoplasia; Penile/Perianal/Perineal Cancer; Anal Cancer; Genital Warts
MeSH Terms: conditions — Anus Neoplasms; Condylomata Acuminata | interventions — Vaccines

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Human Papillomavirus 9-Valent (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) Vaccine (E.coli) (Experimental): Participants in this arm would receive Recombinant Human Papillomavirus 9-Valent (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) Vaccine (E.coli).
  Interventions: Biological: Recombinant Human Papillomavirus 9-Valent (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) Vaccine (E.coli)
- Aluminum Adjuvant (Placebo Comparator): Participants in this arm would receive Aluminum Adjuvant.
  Interventions: Biological: Aluminum Adjuvant

INTERVENTIONS:
Biological: Recombinant Human Papillomavirus 9-Valent (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) Vaccine (E.coli) — Participants received 3 doses of 9-valent HPV vaccine according to a 0, 1, 6-month schedule (0.5 mL intramuscular injection in the deltoid muscle of the upper arm)
  Arms: Recombinant Human Papillomavirus 9-Valent (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) Vaccine (E.coli)
Biological: Aluminum Adjuvant — Participants received 3 doses of Aluminum Adjuvant according to a 0, 1, 6-month schedule (0.5 mL intramuscular injection in the deltoid muscle the upper arm).
  Arms: Aluminum Adjuvant

SUMMARY:
This phase III clinical trial was designed to evaluate the efficacy, immunogenicity and safety of a Recombinant Human Papillomavirus 9-Valent (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) Vaccine (E.Coli) manufactured by Xiamen Innovax Biotech CO., LTD., in Chinese males aged 18-45 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants aged 18-45 years at the time of the first vaccination.
2. Be able to comprehend the trial procedures and comply with the protocol requirements (e.g., providing biological samples, completing diary/contact cards, and attending scheduled follow-up visits), and provide written informed consent.
3. No more than 5 sexual partners so far.
4. Participants who agree to adopt effective contraceptive measures within 30 days after each vaccination.
5. No prior history of HPV-related anal-genital lesions (e.g., genital warts, penile/perineal/perianal intraepithelial neoplasia, penile/perineal/perianal cancer, anal intraepithelial neoplasia, and anal cancer).

Exclusion Criteria:

1. Participants who have received or plan to receive any other HPV vaccine during the study period, or have participated in any other HPV-related clinical trial.
2. Axillary temperature > 37.0°C.
3. Engagement in sexual activity (including vaginal/anal intercourse, or any genital contact) within 48 hours prior to any swab/anal cytology specimen collection visit, or any other behavior that may affect the anal-genital examination and specimen collection (anal procedures only applicable to MSM participants).
4. Presence of clinically vident genital warts, external genital lesions, or anal lesions which may suggest sexually transmitted diseases on the day of enrollment.
5. Participants who received immunosuppressed, immunoregulation therapy or corticosteroid systemic therapy (≥14 consecutive days) within 6 months prior to enrollment, except local treatment (e.g., ointment, eyedrops, inhalants or nasal sprays).
6. Administration of immunoglobulin and/or blood products 3 months prior to vaccination or intending to use them within 7 months after the first dose.
7. Use of any investigational or non-registered product (drug or vaccine) within 30 days prior to vaccination, or intending to use them or participate in another clinical trial during the study period.
8. Administration of inactivated vaccine within 14 days or live vaccine within 21 days before vaccination.
9. Any acute illness requiring systemic antibiotic or antiviral treatment within 5 days prior to vaccination, or axillary temperature ≥38.0°C within 3 days prior to vaccination.
10. A state of immunocompromised condition as inquiried by study investigator, e.g., congenital or acquired immunodeficiency diseases, HIV infection, immune diseases (including systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy, or any other condition that may affect immune response), primary diseases or cancer of major organs (such as heart, liver, spleen, lungs, kidneys).
11. History of severe allergy, including serious adverse reactions (e.g., dyspnea, angioedema) to any previous vaccination, or severe allergy to any component of the trial vaccine (recombinant VLP protein, sodium dihydrogen phosphate, disodium hydrogen phosphate, polysorbate, aluminum hydroxide).
12. Asthma, with unstable condition over the past two years requiring emergency treatment, hospitalization, oral or intravenous corticosteroid administration.
13. History of hypertension or hypotension, not stably controlled despite regular medication, or systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg, or systolic blood pressure <90 mmHg, measured in both arms at rest.
14. History of severe medical conditions (with unstable condition that may require emergency treatment or hospitalization), as inquiried by study investigator.
15. Self-report past coagulation disorders or abnormal coagulation function.
16. Epilepsy, excluding febrile epilepsy under 2 years of age, alcoholic epilepsy 3 years prior to abstinence or simple epilepsy that did not require treatment in the past 3 years.
17. Any medical, psychological, social, occupational, or other condition that may affect the conduct of the clinical trial, according to the investigator's judgment after medical history and physical examination.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9300 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2031-09-30 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58-associated genital warts, Penile/Perineal/Perianal Intraepithelial Neoplasia 1+ (PIN1+), and Penile/Perineal/Perianal cancer (pooled across all specified HPV types) | 0-78 months
  To evaluate the efficacy of the investigational vaccine in preventing HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58-associated genital warts, PIN1+ and Penile/Perineal/Perianal cancer (pooled across all specified HPV types) in the Per-Protocol Set (PPS) population.
HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58-associated Anal Intraepithelial Neoplasia 1+ (AIN1+) and Anal cancer (pooled across all specified HPV types), only in MSM participants | 0-78 months
  To evaluate the efficacy of the investigational vaccine in preventing HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58-associated AIN1+ and Anal cancer in the PPS population of MSM participants.

SECONDARY OUTCOMES:
HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58-related External Genital and Intra-anal 12-month Persistent Infection (pooled across all specified HPV types) | 0-78 months
  To evaluate the efficacy of the investigational vaccine in preventing HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58-related External Genital and Intra-anal 12-month Persistent Infection (pooled across all specified HPV types).
Seroconversion and antibody levels of neutralizing antibodies against HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58 at Month 7 | 0-7 months
  To evaluate the immunogenicity of the investigational vaccine.
Seropositivity and antibody levels of neutralizing antibodies against HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58 at Month 18, 30, 42, 54, 66 and 78 | 18-78 months
  To evaluate the long-term immunopersistence of the investigational vaccine.
Adverse events/reactions occurred within 30 days after each vaccination | Within 30 days (Day 0-30) after each vaccination
  To evaluate the safety of the investigational vaccine.
Serious adverse events occurred throughout the study | 0-78 months
  To evaluate the safety of the investigational vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Master, Study Chair — Xiamen University; Xiaoqiang Liu, Ph.D., Principal Investigator — Yunnan Provincial Center for Disease Control and Prevention; Long Sui, Ph.D., Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University
Locations (4):
- China (4):
  - Fujian Provincial Center for Disease Control and Prevention, Fuzhou, Fujian
  - Sichuan Provincial Center for Disease Control and Prevention, Chengdu, Sichuan
  - Yunnan Provincial Center for Disease Control and Prevention, Kunming, Yunnan
  - Zhejiang Provincial Center for Disease Control and Prevention, Hangzhou, Zhejiang